CLINICAL TRIAL: NCT00702624
Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established After Controlled Ovarian Stimulation in Clinical Trial 107012 for the Development of Org 36286 (Corifollitropin Alfa)
Brief Title: Pregnancy and Neonatal Follow-up of Ongoing Pregnancies Established in Clinical Trial P05690 (Care Program) (P05710)
Acronym: Care
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: P05710; 2006-003812-23 (EudraCT Number); 107014 (Other: Organon); MK-8962-003 (Other: Merck)
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Results first posted 2015-04-30 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy; Neonates
Keywords: Neonatal outcome; Congenital malformations; In-Vitro fertilization; Controlled ovarian stimulation; Follow-up
MeSH Terms: conditions — Congenital Abnormalities | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta; Gonadotropin-Releasing Hormone; Progesterone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Corifollitropin alfa 100 μg: In follow-up study, no medication or investigational product was administered. In base study P05690 (NCT00702845), participants received single subcutaneous (SC) injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo-recombinant Follicle Stimulating Hormone (recFSH) injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants in base study P05690 also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of Human Chorion Gonadotropin (hCG) administration. Participants also received Gonadotropin Releasing Hormone (GnRH) antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day by intramuscular [IM] injection), starting on day of oocyte pick-up (OPU) and continuing for at least 6 weeks or up to menses.
  Interventions: Drug: Corifollitropin alfa; Drug: gonadatropin releasing hormone (GnRH) antagonist ganirelix; Biological: human chorion gonadotropin (hCG); Biological: progesterone; Drug: placebo-recFSH (follitropin beta); Biological: open-label recFSH (follitropin beta)
- recFSH 150 IU: In follow-up study, no medication or investigational product was administered. In base study P05690 (NCT00702845), participants in the reference group received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG (10,000 or 5,000 IU/USP) administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG. Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the day of OPU and continuing for at least 6 weeks or up to menses.
  Interventions: Biological: recFSH (follitropin beta); Drug: gonadatropin releasing hormone (GnRH) antagonist ganirelix; Biological: human chorion gonadotropin (hCG); Biological: progesterone; Drug: placebo-corifollitropin alfa; Biological: open-label recFSH (follitropin beta)

INTERVENTIONS:
Drug: Corifollitropin alfa — Single injection of 100 μg corifollitropin alfa administered under protocol P05690
  Other Names: SCH 900962; MK-8962
  Groups: Corifollitropin alfa 100 μg
Biological: recFSH (follitropin beta) — Daily recFSH administered under protocol P05690
  Other Names: follitropin beta; Puregon®; Follistim®
  Groups: recFSH 150 IU
Drug: gonadatropin releasing hormone (GnRH) antagonist ganirelix — GnRH antagonist ganirelix administered SC at a dose of 0.25 mg/day under protocol P05690
Biological: human chorion gonadotropin (hCG) — hCG 5,000 IU/USP or 10,000 IU/USP administered under protocol P05690
Biological: progesterone — Under protocol P05690, progesterone was started on the day of oocyte pick-up (OPU) and continued for at least 6 weeks or up to menses. Participants received at least 600 mg/day vaginally or 50 mg/day IM.
Drug: placebo-recFSH (follitropin beta) — Placebo-recFSH at the equivalent volume of 150 IU/day administered under protocol P05690
  Groups: Corifollitropin alfa 100 μg
Drug: placebo-corifollitropin alfa — Single SC injection of placebo-corifollitropin alfa on Day 2 or 3 of the menstrual cycle, administered under protocol P05690
  Groups: recFSH 150 IU
Biological: open-label recFSH (follitropin beta) — Open-label recFSH up to a maximum dose of 200 IU/day, administered under protocol P05690

SUMMARY:
The objective of this follow-up study is to evaluate whether corifollitropin alfa (Org 36286) treatment for the induction of multifollicular growth in women undergoing controlled ovarian stimulation (COS) prior to in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) is safe for pregnant participants and their offspring.

DETAILED DESCRIPTION:
This is a follow-up protocol to prospectively monitor pregnancy, delivery, and neonatal outcome of women who were treated with corifollitropin alfa or recFSH and became pregnant during the base study P05690 (NCT00702845). For this trial no study specific assessments are required, but information as obtained in standard practice will be used.

ELIGIBILITY:
Inclusion Criteria:

* Participants who participated in base study P05690 (NCT00702845) and received at least one dose of either corifollitropin alfa (Org 36286) or recFSH in base study P05690;
* Ongoing pregnancy confirmed by ultrasound at least 10 weeks after embryo transfer in base study P05690;
* Able and willing to give written informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with an ongoing pregnancy at least 10 weeks after embryo transfer in base study P05690 (NCT00702845) were enrolled in this trial.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Bonduelle M, Mannaerts B, Leader A, Bergh C, Passier D, Devroey P. Prospective follow-up of 838 fetuses conceived after ovarian stimulation with corifollitropin alfa: comparative and overall neonatal outcome. Hum Reprod. 2012 Jul;27(7):2177-85. doi: 10.1093/humrep/des156. Epub 2012 May 15. PMID 22587997

RESULTS

PARTICIPANT FLOW:
Groups:
- Corifollitropin Alfa 100 μg Women/Expectant Mothers: Participants in base study P05690 received single SC injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo recFSH injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG administration. Participants also received GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP); and progesterone (at least 600 mg/day vaginally or 50 mg/day by intramuscular [IM] injection), starting on day of OPU and continuing at least 6 weeks or up to menses. Eligible participants from base study were enrolled in follow up study P05710, but no study treatments were given.
- recFSH 150 IU Women/Expectant Mothers: Participants in the reference group in base study P05690 received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the Day of hCG administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the Day of OPU and continuing for at least 6 weeks or up to menses. Eligible participants from the base study were enrolled in follow up study P05710, but no study treatments were given.
- Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET: This group includes fetuses of expectant mothers who were administered corifollitropin alfa in base study P05690 (NCT00702845). The fetuses were present at 10 weeks after embryo transfer (ET) in the base study, and expectant mothers were eligible for enrollment in follow up study P05710.
- recFSH 150 IU Fetuses at 10 Weeks After ET: This group includes fetuses of expectant mothers who were administered recFSH on base study P05690 (NCT00702845). The fetuses were present at 10 weeks after ET in the base study, and expectant mothers were eligible for enrollment in follow up study P05710.
Period: Base Study P05690 (NCT00702845)
Arm/Group | Corifollitropin Alfa 100 μg Women/Expectant Mothers | recFSH 150 IU Women/Expectant Mothers | Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET | recFSH 150 IU Fetuses at 10 Weeks After ET
Started | 268 | 128 | 0 | 0
Completed | 246 (To complete study, participants from the base study P05690 (NCT00702845) had embryos transferred.) | 121 (To complete study, participants from the base study P05690 (NCT00702845) had embryos transferred.) | 0 | 0
Not Completed | 22 | 7 | 0 | 0
Period: Expectant Mother Follow-up
Arm/Group | Corifollitropin Alfa 100 μg Women/Expectant Mothers | recFSH 150 IU Women/Expectant Mothers | Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET | recFSH 150 IU Fetuses at 10 Weeks After ET
Started | 68 | 45 | 0 | 0
Completed | 61 (To complete the study, participants must have completed a follow-up visit at 4-12 weeks postpartum.) | 45 (To complete the study, participants must have completed a follow-up visit at 4-12 weeks postpartum.) | 0 | 0
Not Completed | 7 | 0 | 0 | 0
Period: Fetuses/Infant Follow-up
Arm/Group | Corifollitropin Alfa 100 μg Women/Expectant Mothers | recFSH 150 IU Women/Expectant Mothers | Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET | recFSH 150 IU Fetuses at 10 Weeks After ET
Started | 0 | 0 | 88 | 55
Live Born Infants | 0 | 0 | 80 (Infants born to eligible mothers were followed for safety and efficacy) | 55 (Infants born to eligible mothers were followed for safety and efficacy.)
Completed | 0 | 0 | 78 (To complete the study, infants must have completed a follow-up visit at 4-12 weeks postpartum.) | 55 (To complete the study, infants must have completed a follow-up visit at 4-12 weeks postpartum.)
Not Completed | 0 | 0 | 10 | 0

BASELINE CHARACTERISTICS:
Population: Individuals who participated in base study P05690 (NCT00702845) and received at least one dose of either corifollitropin alfa or recFSH, who had an ongoing pregnancy confirmed by ultrasound at least 10 weeks after ET in base study P05690 and were able and willing to give written informed consent.
Groups:
- Corifollitropin Alfa 100 μg Expectant Mothers: Participants in base study P05690 received single SC injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo recFSH injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG administration. Participants also received GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP); and progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on day of OPU and continuing at least 6 weeks or up to menses. Eligible participants from base study were enrolled in follow up study P05710, but no study treatments were given.
- recFSH 150 IU Expectant Mothers: Participants in the reference group in base study P05690 received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the Day of hCG administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the Day of OPU and continuing for at least 6 weeks or up to menses. Eligible participants from the base study were enrolled in follow up study P05710, but no study treatments were given.
- Total: Total of all reporting groups
Arm/Group | Corifollitropin Alfa 100 μg Expectant Mothers | recFSH 150 IU Expectant Mothers | Total
Number analyzed (Participants) | 68 | 45 | 113
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (3.3) | 31.3 (3.1) | 30.8 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 45 | 113
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With ≥1 Live Born Infant During Follow-up (Take-Home Baby Rate)
Description: The Take-Home Baby Rate was defined as the number of participants with an ongoing pregnancy in base study P05690 with at least one live born infant during follow up relative to the number of participants treated in base study.
Time Frame: From approximately 10 weeks after ET in base study P05690 up to birth of infant (up to approximately 6 months)
Population: Intent-to-Treat (ITT) group from base study P05690 (NCT00702845), which consisted of randomized participants who were treated with corifollitropin alfa or recFSH.
Measure: Number; unit: Percentage of participants
Groups:
- Corifollitropin Alfa 100 μg Women: Participants in base study P05690 received single SC injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo recFSH injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG administration. Participants also received GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP); and progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on day of OPU and continuing at least 6 weeks or up to menses. Eligible participants from base study were enrolled in follow up study P05710, but no study treatments were given.
- recFSH 150 IU Women: Participants in the reference group in base study P05690 received a single SC injection of placebo-corifollitropin alfa administered on Day 2 or 3 of the menstrual cycle and daily SC recFSH 150 IU injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants also received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including the Day of hCG administration. Participants also received the GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including the Day of hCG (10,000 or 5,000 IU/USP). Participants also received progesterone (at least 600 mg/day vaginally or 50 mg/day IM), starting on the Day of OPU and continuing for at least 6 weeks or up to menses. Eligible participants from the base study were enrolled in follow up study P05710, but no study treatments were given.
Arm/Group | Corifollitropin Alfa 100 μg Women | recFSH 150 IU Women
Number analyzed (Participants) | 268 | 128
Percentage of participants | 23.5 | 34.4

2. Primary Outcome: Number of Expectant Mothers Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From approximately 10 weeks after ET in base study P05690 up to birth of infant (up to approximately 6 months)
Population: Follow-up safety analysis was performed on expectant mothers who received corifollitropin alfa or recFSH on base study P05690 (NCT00702845) and who enrolled on the follow-up study.
Measure: Number; unit: Participants
Arm/Group | Corifollitropin Alfa 100 μg Expectant Mothers | recFSH 150 IU Expectant Mothers
Number analyzed (Participants) | 68 | 45
Participants | 48 | 35

3. Primary Outcome: Number of Expectant Mothers Experiencing Serious AEs (SAEs)
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect.
Time Frame: From approximately 10 weeks after ET in base study P05690 up to birth of infant (up to approximately 6 months)
Population: as for outcome 2
Measure: Number; unit: Participants
Groups:
- Corifollitropin Alfa 100 μg Expectant Mothers: Participants in base study P05690 received single SC injection of corifollitropin alfa 100 μg (Org 36286) on Day 2 or 3 of menstrual cycle and daily placebo recFSH injections (7 total) from Stimulation Day 1 up to and including Stimulation Day 7. Participants received open-label recFSH (up to 200 IU/day) from Stimulation Day 8 onwards, up to and including Day of hCG administration. Participants also received GnRH antagonist ganirelix (0.25 mg) once daily SC starting on Stimulation Day 5 up to and including Day of hCG (10,000 or 5,000 IU/USP); and progesterone (at least 600 mg/day vaginally or 50 mg/day by intramuscular [IM] injection), starting on day of OPU and continuing at least 6 weeks or up to menses. Eligible participants from base study were enrolled in follow up study P05710, but no study treatments were given.
Arm/Group | Corifollitropin Alfa 100 μg Expectant Mothers | recFSH 150 IU Expectant Mothers
Number analyzed (Participants) | 68 | 45
Participants | 38 | 21

4. Primary Outcome: Number of Infants Experiencing AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to 12 weeks after birth
Population: Follow-up safety analysis was performed on live born infants delivered by expectant mothers who received corifollitropin alfa or recFSH on base study P05690 (NCT00702845) and who enrolled on the follow-up study.
Measure: Number; unit: Live born infants
Groups:
- Corifollitropin Alfa 100 μg Follow-Up Infants: Infants that were born to eligible mothers who received SC corifollitropin alfa plus hCG on base study P05690 (NCT00702845) were followed for safety and efficacy on the current follow-up study (P05710) according to standard practice.
- recFSH 150 IU Follow-Up Infants: Infants that were born to eligible mothers who received SC recFSH plus hCG on base study P05690 (NCT00702845) were followed for safety and efficacy on the current follow-up study (P05710) according to standard practice.
Arm/Group | Corifollitropin Alfa 100 μg Follow-Up Infants | recFSH 150 IU Follow-Up Infants
Number analyzed (Participants) | 80 | 55
Live born infants | 37 | 27

5. Primary Outcome: Number of Infants Experiencing SAEs
Description: as for outcome 3
Time Frame: Up to 12 weeks after birth
Population: as for outcome 4
Measure: Number; unit: Live born infants
Arm/Group | Corifollitropin Alfa 100 μg Follow-Up Infants | recFSH 150 IU Follow-Up Infants
Number analyzed (Participants) | 80 | 55
Live born infants | 30 | 16

ADVERSE EVENTS:
Time Frame: From approximately 10 weeks after ET in base study P05690 (NCT00702845) up to 12 weeks after birth in current follow-up study (up to approximately 9 months)
Arm/Group | Corifollitropin Alfa 100 μg Expectant Mothers | recFSH 150 IU Expectant Mothers | Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET | recFSH 150 IU Fetuses at 10 Weeks After ET
Serious Adverse Events (participants affected / at risk) | 38/68 | 21/45 | 31/88 | 16/55
Other Adverse Events (participants affected / at risk) | 13/68 | 17/45 | 9/88 | 5/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 100 μg Expectant Mothers (N=68) | recFSH 150 IU Expectant Mothers (N=45) | Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET (N=88) | recFSH 150 IU Fetuses at 10 Weeks After ET (N=55)
Mitral valve prolapse (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia foetal (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia foetal (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intrauterine infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cervix dystocia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Complication of delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal macrosomia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal malposition (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pregnancy induced hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 5 (5) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 4 (4) | 0 (0) | 0 (0)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 3 (3) | 0 (0) | 0 (0)
Uterine contractions during pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Uterine hypotonus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervix cerclage procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aplasia cutis congenita (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Congenital infection (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital pneumonia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Congenital pulmonary artery anomaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital pyelocaliectasis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Congenital syphilis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pulmonary artery stenosis congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinopathy of prematurity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever neonatal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema neonatal (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 8 (8) | 6 (6)
Neonatal cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur functional (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction foetal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 20 (20) | 9 (9)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
Nephrocalcinosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoventilation neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infantile apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 100 μg Expectant Mothers (N=68) | recFSH 150 IU Expectant Mothers (N=45) | Corifollitropin Alfa 100 μg Fetuses at 10 Weeks After ET (N=88) | recFSH 150 IU Fetuses at 10 Weeks After ET (N=55)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 0 (0) | 2 (2)
Abnormal labour (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (2)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (6) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by the Sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in this protocol will first be submitted to Sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.